CLINICAL TRIAL: NCT06322368
Title: Effects of a Combined Myofunctional and Respiratory Intervention on Phonation in Patients With Chronic Stroke
Brief Title: Myofunctional and Respiratory Intervention on Phonation in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Cabrera Martos, Profesor titular de Universidad, Universidad de Granada
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF002
Record Dates: First submitted 2024-01-31; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Range of Motion, Articular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofunctional and respiratory training (Experimental): Patients with chronic stroke receiving an exercise training program for the muscles around the face, mouth, and tongue and a respiratory training focused on inspiratory and expiratory muscle strengthening.
  Interventions: Other: Myofunctional and respiratory training program
- Range of motion and stimulation exercises (Active Comparator): Standard treatment focused mainly on range of motion, such as opening and closing the mouth and stimulation exercises
  Interventions: Other: Range of motion and thermal and mechanical stimulation exercising

INTERVENTIONS:
Other: Myofunctional and respiratory training program — The patients will receive exercises included in a myofunctional approach and a respiratory training focused on inspiratory and expiratory muscles using a device.
  Arms: Myofunctional and respiratory training
Other: Range of motion and thermal and mechanical stimulation exercising — The patients will receive the standard treatment of speech and language therapy including range of motion exercises (open and close the mouth) and thermal and mechanical stimulation in the orofacial region.
  Arms: Range of motion and stimulation exercises

SUMMARY:
Patients with stroke frequently present phonation difficulties. An intervention combining myofunctional and respiratory training is presented in order to improve phonation outcomes.

DETAILED DESCRIPTION:
Patients with stroke frequently present phonation difficulties. An intervention combining myofunctional and respiratory training is presented to improve phonation outcomes. Myofunctional therapy is based on exercise training program for the muscles around your face, mouth, and tongue. Respiratory muscle strength training focuses on increasing the force-generating capacity of the inspiratory and expiratory muscles. A combination of both may be of interest to improve phonation parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of chronic stroke (duration above 6 months).
* Age over 18 years

Exclusion Criteria:

* Communication or cognitive deficits that prevented them from following verbal commands.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Volume during monologue | Baseline, 6 weeks
  The volumen during a monologue of basic activities of daily living assessed in decibels.
Frequency during monologue | Baseline, 6 weeks
  The frequency during a monologue of basic activities of daily living expressed in hertz.

SECONDARY OUTCOMES:
Volumen during sustained phonation of /s/ sound | Baseline, 6 weeks
  The decibels during the maximum sustained phonation of s.
Communication effectiveness Index | Baseline, 6 weeks
  This is a questionnaire with the scores ranging from 0 to 100, with lower scores meaning more difficulties associated to effectiveness in communication.
Frequency during sustained phonation of /s/ sound | Baseline, 6 weeks
  The Hertzs during the maximum sustained phonation of s.
Volumen during sustained phonation of /a/ sound | Baseline, 6 weeks
  The decibels during the maximum sustained phonation of a.
Frequency during sustained phonation of /a/ sound | Baseline, 6 weeks
  The Hertzs during the maximum sustained phonation of a

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cabrera Martos, Principal Investigator — UGR
Locations (1):
- Faculty of Health Sciences, Granada, Spain

IPD SHARING:
Plan to Share IPD: No